CLINICAL TRIAL: NCT03616678
Title: Evaluation of The Minimally Invasive VenTouch™ System in The Treatment of Functional Mitral Valve Regurgitation (FMR): OUS Feasibility Study
Brief Title: VenTouch OUS Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mardil Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VenTouch CT007
Record Dates: First submitted 2018-07-24; First posted 2018-08-06 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Functional Mitral Regurgitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VenTouch System Implant (Experimental): The VenTouch System is intended for use in the treatment of functional MR (FMR) in adults who are symptomatic despite optimal medical management. It is indicated for subjects with FMR with essentially normal leaflet anatomy and motion, with mitral valve regurgitation attributable to annular and/or ventricular dilation. It is not intended to treat structural defects/degeneration of the mitral valve. The VenTouch System is intended to provide ventricular support that will encourage beneficial remodeling of the heart and, with adjustable inflatable chambers, it is intended to reduce annular dilation, correct papillary muscle displacement, and restore mitral valve leaflet coaptation, allowing proper closure of the valve, and reducing or eliminating MR. The VenTouch System is indicated for patients who have "moderately severe" or "severe" mitral regurgitation (grade 3 or 4 MR).
  Interventions: Device: VenTouch System

INTERVENTIONS:
Device: VenTouch System — The VenTouch™ System consists of a delivery tool with a pre-loaded implant (VenTouch device) and accessories, which include a sizing tool, PEMS, chamber positioning tool, and accessories kit with luer fitting, tubing clamp, and titanium plug. The VenTouch device is offered in 6 sizes, with 4 different sized inflatable chambers available. Please refer to the VenTouch Instructions for Use for and system details.
  The VenTouch device consists of three (3) inflatable silicone chambers attached to the wall of a knitted polyester support. The VenTouch device is implanted around the base of the heart and positioned at the level of the atrio-ventricular (AV) groove and the adjacent ventricular muscle. The VenTouch device is composed of biocompatible, medical-grade silicone and polyester.

SUMMARY:
This is a prospective, multi-center, single-arm study to evaluate safety and efficacy of the VenTouch System for treatment of subjects with functional MR.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm study to evaluate safety and efficacy of the VenTouch System for treatment of subjects with functional MR enrolling up to 15 subjects who have been diagnosed with Grade 3-4 functional mitral valve regurgitation and deemed eligible per assessment by the inclusion/exclusion criteria. The duration of the study follow-up is 36 months from the time of therapy adjustment. Data from this trial may be utilized in support of a CE study in Europe and/or a pilot IDE study in the U.S. Follow-up testing will be performed at 1, 3, 6, 12, 24, and 36 months post-therapy adjustment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age
2. Symptomatic FMR of grade moderately severe to severe (3 to 4) due to either ischemic or non-ischemic dilated cardiomyopathy with structurally normal leaflets determined by echocardiography (preferably with echocardiographic evidence of EROA ≥ 0.20 cm2)
3. NYHA Class II to IV
4. Left Ventricular Ejection Fraction (LVEF) 20%-50% determined by echocardiography
5. Treatment and compliance with optimal guideline-directed medical therapy for heart failure for at least 30 days
6. Subjects with a Class I indication for CRT implant according to current guidelines should have CRT implant prior to entry into the study. Subjects who have existing CRT implants may be included in the study if the implant has been in place for at least 90 days; reprogramming of an implanted CRT that results in increased biventricular pacing (from <92% to ≥92%) must be in place for at least 30 days.
7. Left Ventricular End Diastolic Diameter (LVEDD) of 55 to 80 mm as determined by echocardiography
8. Indexed Left Ventricular End Diastolic Diameter (LVEDDi) of 30 to 40 mm/m2 (where LVEDDi is calculated by LVEDD/Body Surface Area (BSA))
9. Subject is willing and available to return for study follow-up
10. Subject or legal representative understands and provides signed informed consent for participation in study
11. Acceptance of subject for trial enrollment after review of all subject baseline data by Study Selection Committee

Exclusion Criteria:

1. Life expectancy of less than 12 months due to conditions other than cardiac status
2. Anticipated need for LVAD or transplant within 12 months
3. Chronic Obstructive Pulmonary Disease (COPD) requiring continuous home oxygen therapy or chronic outpatient oral steroid use
4. American College of Cardiology / American Heart Association (ACC/AHA) Stage D heart failure
5. Six-minute walk distance < 150 meters
6. Identified need for any cardiovascular surgery
7. STS score that suggests prohibitive surgical risk as determined by Subject Selection Committee
8. Untreated clinically significant coronary artery disease
9. Any procedure, condition or cardiac anatomy that may impact or compromise the pericardial space (e.g. prior mitral valve surgery, CABG, epicardial pacing leads, pericarditis, or other procedure involving pericardial access)
10. Percutaneous coronary intervention, acute coronary syndrome (e.g. STEMI or non-STEMI myocardial infarction, unstable angina) or clinically significant cardiac events (e.g. hypotension, syncope, arrhythmias, embolism, heart failure exacerbation or any hospitalization) within 30 days of enrollment
11. Thoracic or cardiac surgery contraindication (e.g., acute respiratory distress, endocarditis, myocarditis, pericarditis)
12. Significant structural abnormality of the mitral valve (e.g. flail leaflets, ruptured or elongated chordae, prolapsed valve, perforated valve leaflets, significant calcification in the annulus, or calcification in the leaflets that restricts motion)
13. Severe symptomatic carotid stenosis
14. Severe or sustained pulmonary hypertension, defined by resting pulmonary artery systolic (PAS) pressure ≥70 mmHg determined by echocardiography or right heart catheterization
15. Physical evidence of right-sided congestive heart failure with echocardiographic evidence of moderate or severe right ventricular dysfunction or moderate to severe TR
16. Hypotension (systolic pressure <90 mmHg)
17. Hemodynamic instability requiring inotropic support or mechanical heart assistance within 30 days
18. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, or any other structural heart disease causing heart failure other than dilated cardiomyopathy
19. UNOS status 1 heart transplantation
20. Creatinine > 2.5 mg/dL (221 µmol/L) and/or renal failure requiring dialysis
21. Stroke (cerebrovascular accident) or transient ischemic event (TIA) within 30 days of enrollment
22. Active systemic infection or bleeding
23. Autoimmune disorders and/or the use of immune suppression therapy
24. Females who are pregnant (as documented by HCG beta pregnancy test in females of child-bearing age) or lactating
25. Currently enrolled in another investigational drug or device study

Intra-Operative Exclusion Criteria:

1. Significant structural abnormality of the mitral valve (e.g. flail leaflets, ruptured or elongated chordae, prolapsed valve, perforated valve leaflets, significant calcification in the annulus, or calcification in the leaflets that restricts motion)
2. Signs/indications of ischemia
3. Intra-operative coronary angiography demonstrates that there is compression of the coronary arteries or reduction in coronary blood flow due to the VenTouch implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate procedural feasibility through successful completion of implant and therapy adjustment procedures | Intra-operative
  Evaluate procedural feasibility through successful completion of implant and therapy adjustment procedures and intraoperative transesophageal echocardiographic (TEE) evidence of MR severity reduction (a minimum of one grade)
Evaluate SAE Rates | 1 Month
  Evaluate Serious Adverse Event (SAE) rates at 1 month post-therapy adjustment

SECONDARY OUTCOMES:
Evaluate SAE Rates | 36 Months
  Evaluate Serious Adverse Event (SAE) rates
Evaluate MR Severity | 36 Months
  Evaluate MR severity reduction and mitral valve dimension reduction via echocardiographic core lab assessment
Evaluate Reverse Ventricular Remodeling | 36 Months
  Evaluate reverse ventricular remodeling via echocardiographic core lab assessment
Evaluate Changes in Patient Symptoms by NYHA | 36 Months
  Evaluate changes in patient symptoms as assessed by the NYHA functional class
Evaluate Changes in Patient Functional Status by Six-Minute Walk | 36 Months
  Evaluate changes in patient functional status as assessed by Six-Minute Walk
Evaluate Changes in Patient Functional Status by KCCQ | 36 Months
  Evaluate changes in patient functional status as assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ)

CONTACTS AND LOCATIONS:
Locations (12):
- Canada (6):
  - Libin Cardiovascular Institute, University of Calgary, Calgary, Alberta
  - University of British Columbia, St. Paul's Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, University Hospital, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie De Québec (IUCPQ), Québec, Quebec
- Bordeaux Heart University Hospital, Bordeaux, Pessac, France
- CardioVasculäres Centrum, Frankfurt, Germany
- Semmelweis University Heart and Vascular Center, Budapest, Hungary
- Leiden University Medical Center, Leiden, Netherlands
- Pacifica Salud Hospital Punta Pacifica, Panama City, Panama
- Centralny Szpital Kliniczny MSWiA w Warszawia, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Sponsor Website — http://www.mardil.com